CLINICAL TRIAL: NCT02651441
Title: Randomized, Controlled Study of the Safety and Efficacy of D-CIK Immune Cell Combined With Chemotherapy for Non-Small Cell Lung Cancer
Brief Title: D-CIK Combined With Chemotherapy for Non-Small Cell Lung Cancer(NSCLC)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Hornetcorn Bio-technology Company, LTD (Industry)
Collaborators: Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HYK-NSCLC
Record Dates: First submitted 2016-01-05; First posted 2016-01-11 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-01

CONDITIONS: Lung Cancer; Non-small Cell Lung Cancer
Keywords: D-CIK; lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- D-CIK (Experimental): After accepting chemotherapy of Gemcitabine and Cisplatin according to NCCN guidelines,patients will receive 3 cycles of D-CIK treatment.
  Interventions: Drug: Gemcitabine; Drug: Cisplatin; Biological: D-CIK
- Chemotherapy (Active Comparator): After accepting chemotherapy of Gemcitabine and Cisplatin according to NCCN guidelines, patients will just regularly follow up.
  Interventions: Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine 1000mg/m2 IV on day1 and day8, repeat every 3 weeks.
  Other Names: Gemzar
Drug: Cisplatin — Cisplatin 25mg/m2 IV on day 1,2 and 3, repeat every 3 weeks.
  Other Names: cisplatinum
Biological: D-CIK — 8×10^9 D-CIK cells for each infusion, IV (in the vein) for 3 cycles, each cycle received four infusions on day 14, 16, 30 and 32.
  Arms: D-CIK

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of chemotherapy combined with dendritic activated cytokine-induced killer cell (D-CIK) for non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
60 patients with stage Ⅲb～Ⅳ NSCLC will be randomly divided into group A（receive D-CIK treatment and chemotherapy) or group B（just receive chemotherapy),and the randomize ratio will be 1:1. Patients in group A will receive 3 cycles of D-CIK treatment (every 1 months) and 4 cycles of chemotherapy (every 2 weeks).Patients in group B will receive only 4 cycles chemotherapy（every 2 weeks).

ELIGIBILITY:
Inclusion Criteria:

* The patient who have singed the informed consent;
* Histologically confirmed with NSCLC at stage Ⅲb～Ⅳ;
* Expected survival time is more than 2 month;
* Eastern Cooperative Oncology Group (ECOG) performance status was 0-2.

Exclusion Criteria:

* Hemoglobin<8.0 g/dL,White blood cell <3 x 10^9/L;Platelet count <75 x 10^9/L; ALT, AST, BUN and Cr more than normal limits on 3.0 times;
* Known or suspected allergy to the investigational agent or any agent given in association with this trial;
* Pregnant or lactating patients;
* Known history of Human Immunodeficiency Virus (HIV), Hepatitis C Virus (HCV) or TreponemaPallidun (TP) infection;
* Patients who are suffering from serious autoimmune disease;
* Patients who had used long time or are using immunosuppressant;
* Patients who had active infection;
* Patients who are suffering from serious organ dysfunction;
* Patients who are suffering from other cancer;
* Other situations that the researchers considered unsuitable for this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-02; Primary Completion 2019-05 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Progress-free survival | 3 years

SECONDARY OUTCOMES:
Overall survival | 3 years
Quality of life (QOL) | 3 years
  The assessment will be performed using The European Organization for Research and Treatment of Cancer QLQ-C30 (EORTC-QLQ-C30).
Phenotypic analysis of T cells | 1 year
  The number of CD3+ (or CD8+ or CD4+ or CD56+) T cell
Severity of adverse events | 1 year
  According to National Cancer Institute Common Terminology Criteria for Adverse Events（NCI-CTCAE)

CONTACTS AND LOCATIONS:
Overall Officials: Zhi Z Zhang, Professor, Principal Investigator — Affiliated Tumor Hospital of Guangzhou Medical University immunotherapy center
Locations (1):
- Affiliated Tumor Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided